CLINICAL TRIAL: NCT04420624
Title: COLchicine to Prevent Sympathetic Denervation After an Acute Myocardial Infarction
Acronym: COLD-MI
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Inclusion period completed
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RECHMPL18_0459; 2020-000098-25 (Registry Identifier: EudraCT)
Record Dates: First submitted 2020-04-29; First posted 2020-06-09 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2022-12

CONDITIONS: Myocardial Infarction, Acute
Keywords: Myocardial infarction; Sympathetic denervation; Heart failure
MeSH Terms: conditions — Myocardial Infarction; Heart Failure | interventions — Colchicine

STUDY DESIGN:
Intervention Model Description: Prospective, phase IIb, monocentric, randomized, open labeled with 2 parallel study arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Colchicine (Experimental): colchicine and standard therapy
  Interventions: Drug: Colchicine
- Comparator (No Intervention): standard therapy

INTERVENTIONS:
Drug: Colchicine — 1 mg (or 0.5mg) tablet of colchicine taken once a day for 1 month
  Other Names: no other name
  Arms: Colchicine

SUMMARY:
This study evaluates the benefit of colchicine on induced denervation after myocardial infarction. Patients who have suffered a documented De Novo myocardial infarction and completed a revascularization procedure will receive either colchicine on top of standard therapy, compared to standard therapy alone (1:1 allocation ratio). Colchicine 1mg (or 0.5mg) will be initiated within 48h after percutaneous revascularization and prescribed for one month.

DETAILED DESCRIPTION:
COLD-MI study aims to explore colchicine's impact on myocardial denervation following reperfused acute myocardial infarction. Acute myocardial infarction is the leading cause of heart failure (HF). It induces myocardial denervation predisposing to ventricular rhythm disorders and death. This denervation linked to infarction's size occurs by direct ischaemic mechanisms during the initial coronary occlusion (initially non-vascularised zone) and secondarily by cardiac remodelling in the context of the heart failure (HF). In usual practice, cardiac denervation which intensity is correlated with rhythm and mortality risks, can be evaluated by scintigraphy. In a murine reperfusion model of ischemia, the direct anti-inflammatory effect of colchicine reduces the size of the necrosis and improves post-ischemic remodeling. This suggests that colchicine may reduce myocardial denervation.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 80 year old
* Hospitalization within 12 hours of onset of acute chest pain
* Patient must have suffered a documented acute myocardial infarction
* Coronary occlusion on initial angiography (culprit artery with aTIMI (Thrombolysis in Myocardial Infarction) flow 1 or 0)
* Patient eligible for a revascularization procedure by PTCA (Percutaneous transluminal coronary angioplasty)

Exclusion Criteria:

* Patients with a history of myocardial infarction prior to the current episode
* Patient in cardiogenic shock or with hemodynamic instability
* Patients with severe hepatic or renal dysfunction (GFR ≤30 mL/min)
* Pregnant women or women of childbearing age without contraception
* Treatment with a potent CYP3A4 inhibitor or a P-glycoprotein inhibitor in patients with renal or hepatic impairement
* Association with macrolides (except spiramycin)
* Association with pristinamycin

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-12-04 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-05-24 (Actual)

PRIMARY OUTCOMES:
Percentage of myocardial denervation | 6 month
  assess by MIBG (méta-iodobenzylguanidine)-nuclear cardiac imaging

SECONDARY OUTCOMES:
Change in the heart-to-mediastinum ratio | 6 month
  The heart-to-mediastinum (H/M) ratio, the heart count normalized for the mediastinum count, is used as a quantitative index in cardiac 123 I-MIBG imaging.
Left Ventricular Ejection Fraction in percent | 6 month
  By transthoracic echocardiogram (TTE)
Left Ventricular Ejection Fraction in percent | 6 month
  By MIBG (méta-iodobenzylguanidine)-nuclear cardiac imaging
Left Ventricular Ejection Fraction in percent | 1 month
  By transthoracic echocardiogram (TTE)
Change in Sinus variability | 6 month
  by 24 hours holter recording : SDNN (Standard Deviation of NN intervals) will be measured
Change in Sinus variability | 1 month
  by 24 hours holter recording : SDNN (Standard Deviation of NN intervals) will be measured
Basic ECG parameters (QRS duration) | 6 month
Basic ECG parameters (QRS duration) | 1 month
Basic ECG parameters (corrected QT) | 1 month
Basic ECG parameters (corrected QT) | 6 month
Number of ventricular extrasystole (2 or 3 VES) per 24 hours on the Holter | 6 month
Number of bursts (2 or 3 VES) per 24 hours on the Holter | 1 month
Number of bursts (2 or 3 VES) per 24 hours on the Holter | 6 month
Number of ventricular or supraventricular tachycardia (>3 VES) episodes per 24 hours | 1 month
Number of ventricular or supraventricular tachycardia (>3 VES) episodes per 24 hours | 6 month
Time from randomization to death (total mortality) | 6 month
Time from randomization to heart failure hospitalization | 6 month
Time from randomization to all-cause hospitalization | 6 month
Variations in the levels of neurotrophic molecular markers | Between hospitalization and 1 month
  Concentration of NGF ng/mL
Variations in the levels of neurotrophic molecular markers | Between 1 month and 6 months
  Concentration of NGF ng/mL
Variations in the levels of neurotrophic molecular markers | Between hospitalization and 1 month
  Concentration of proNGF ng/mL
Variations in the levels of neurotrophic molecular markers | Between 1 month and 6 months
  Concentration of proNGF ng/mL
Variations in the levels of neurotrophic molecular markers | Between hospitalization and 1 month
  Concentration of BDNF ng/mL
Variations in the levels of neurotrophic molecular markers | Between 1 month and 6 months
  Concentration of BDNF ng/mL
Biological evaluation of infarction size Creatine PhosphoKinase (CPK) | During hospitalization (Day 1 to Day 5)
  Area Under Curve (AUC) of CPK
Biological evaluation of infarction size (troponin) | During hospitalization (Day 1 to Day 5)
  Area Under Curve (AUC) of Troponin
Post infarction systemic inflammation evaluation | Between hospitalization and 1 month
  Concentration of biomarkers from blood : CRP (mg/L)
Post infarction systemic inflammation evaluation | Between 1 month and 6 months
  Concentration of biomarkers from blood : CRP (mg/L)
Post infarction systemic inflammation evaluation | Between hospitalization and 1 month
  Concentration of biomarkers from blood : sST2 (ng/mL)
Post infarction systemic inflammation evaluation | Between 1 month and 6 months
  Concentration of biomarkers from blood : sST2 (ng/mL)
Infarct size in percentage of left ventricular | 6 month
Number of Adverse event | from randomization to 6 months
  Comparison of adverse events between 2 arms

CONTACTS AND LOCATIONS:
Locations (1):
- UH Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No